CLINICAL TRIAL: NCT06922318
Title: A Phase II Study of Sequential Bipolar Androgen Therapy and ZEN-3694 in Sequence With Enzalutamide + ZEN-3694 in Asymptomatic Patients With Metastatic CRPC: The COSMYC Trial (COmbined Suppression of MYC)
Brief Title: The COSMYC Trial (COmbined Suppression of MYC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Zenith Epigenetics (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J2513; IRB00480365 (Other: JHM IRB); P50CA272391 (NIH)
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate Cancer; ZEN-3694; Bipolar androgen therapy; testosterone cypionate; enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — testosterone 17 beta-cypionate; enzalutamide; Gonadotropin-Releasing Hormone; Goserelin; Triptorelin Pamoate; luprolide acetate gel depot; Leuprolide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BATZEN (Experimental): ZEN-3694 48 mg (one 48 mg tablet) will be taken once per day by mouth each cycle (each cycle is 28 days). On the first day of each cycle, testosterone cypionate (400 mg) injection will be administered into the buttocks. The participant will continue with additional 28-day cycles of ZEN-3694 pills and testosterone injections until there is disease progression on bone and CT scans.
  Interventions: Drug: ZEN-3694; Drug: Testosterone cypionate; Drug: Luteinizing hormone-releasing hormone (LHRH) analogue
- ZENZA (Experimental): ZENZA cycles will begin once there is disease progression on bone and CT scans.ZEN-3694 dose will increase to 72 mg (one 48 mg and two 12 mg tablets) to be taken daily by mouth. Enzalutamide 160 mg (four 40 mg capsules) will be taken daily by mouth.
  Interventions: Drug: ZEN-3694; Drug: Enzalutamide; Drug: Luteinizing hormone-releasing hormone (LHRH) analogue

INTERVENTIONS:
Drug: ZEN-3694 — One ZEN-3694 pill (48 mg) will be taken each day of each BATZEN cycle.
Drug: Testosterone cypionate — On day 1 of each BATZEN cycle testosterone cypionate (400 mg) injection to the buttocks will be administered.
  Arms: BATZEN
Drug: Enzalutamide — Enzalutamide 160 mg (four 40 mg capsules) taken daily by mouth on each ZENZA cycle.
  Arms: ZENZA
Drug: Luteinizing hormone-releasing hormone (LHRH) analogue — Patients will continue on ADT with LHRH agonist (i.e. Zoladex, Trelstar, Eligard or Lupron) or LHRH antagonist (Degarelix or Relugolix) if not surgically castrated throughout the duration of the study to inhibit endogenous testosterone production.
  Other Names: Zoladex; Trelstar; Eligard; Lupron; Degarelix; Relugolix

SUMMARY:
This research is being done to determine if receiving the combination of testosterone and ZEN-3694 followed by the combination of enzalutamide plus ZEN-3694 will decrease the size of tumors in patients with prostate cancer that has become resistant to castration and other therapies. The investigators also want to determine if dosing first with the combination of testosterone and ZEN-3694 may cause enzalutamide and ZEN-3694 to work more effectively.

DETAILED DESCRIPTION:
The primary objectives of the study are first to determine if treatment with the combination of ZEN-3694 and Bipolar Androgen Therapy (i.e. BATZEN) will improve the progression-free survival in patients with metastatic castrate-resistant prostate cancer (mCRPC) compared with historical controls. The second primary objective is to determine if treatment with ZEN-3694 and Enzalutamide (i.e. ZENZA) after progression on Bipolar Androgen Therapy (BAT) will improve PSA-progression-free survival compared to historical controls.

Asymptomatic patients with mCRPC without pain due to prostate cancer will be treated on an open label study to evaluate effectiveness of sequential treatment with the combination of ZEN-3694 and high dose testosterone in sequence with enzalutamide and ZEN-3694 to improve primary and secondary outcomes.

Eligible patients are those with mCRPC who have progressive disease after treatment with a second-generation AR-axis inhibitor (Abiraterone, Enzalutamide, Darolutamide, or Apalutamide) used as treatment for castration-sensitive or castration-resistant disease. Patients will continue on Androgen Deprivation Therapy (ADT) with LHRH agonist (i.e. Zoladex, Trelstar, Eligard, or Lupron) or LHRH antagonist (Degarelix or Relugolix) if not surgically castrated throughout the duration of the study to inhibit endogenous testosterone production. One cycle of treatment will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance status ≤2.
2. Age ≥18 years.
3. Histologically-confirmed adenocarcinoma of the prostate.
4. Treated with continuous androgen ablative therapy (either surgical castration or LHRH agonist/antagonist).
5. Documented castrate level of serum testosterone (<50 ng/dl).
6. Metastatic disease radiographically documented by CT or bone scan. While CT scan is preferred, Prostate-Specific Membrane Antigen (PSMA) scan (e.g. Pylarify) may be substitute for CT scan if evidence of metastatic disease observed on the CT portion of the PSMA scan.
7. Must have had disease progression while on a second-generation AR-axis inhibitor (Abiraterone, Enzalutamide, Darolutamide, or Apalutamide) based on:

   PSA progression defined as an increase in PSA, as determined by 2 separate measurements taken at least 1 week apart i. And/ Or Radiographic disease progression, based on RECIST 1.1 in patients with measurable soft tissue lesions or PCWG3 for patients with bone disease
8. Screening PSA must be ≥ 1.0 ng/mL.
9. Patients with soft tissue lesion amenable to biopsy must agree to biopsy collection pre-treatment and at a defined point on treatment to perform tumor tissue analysis.
10. Prior treatment with Provenge vaccine, 223 Radium (Xofigo), poly(ADP-ribose) polymerase (PARP) inhibitors, taxane chemotherapy, Pluvicto, antiandrogens (including enzalutamide, darolutamide, and apalutamide), and radiation is allowed if >4 weeks from last dose.
11. Prior treatment with BAT is allowed if the patient has progressed on an AR-axis inhibitor (i.e. abiraterone or antiandrogen) since BAT treatment.
12. Patients must be withdrawn from second-generation AR-axis inhibitor (Abiraterone, Enzalutamide, Darolutamide, or Apalutamide) for ≥ 2 weeks.
13. Attempts must be made to wean patients off prednisone prior to starting therapy. Patients who cannot be weaned due to symptoms may continue on lowest dose of prednisone achieved during weaning period.
14. Acceptable liver function:

    1. Bilirubin < 2.5 times institutional upper limit of normal (ULN)
    2. Aspartate Transferase (AST) (SGOT) and Alanine Transaminase (ALT) (SGPT) < 2.5 times ULN
15. Acceptable renal function:

    a. Serum creatinine <2.5 times ULN
16. Acceptable hematologic status:

    1. Absolute neutrophil count (ANC) ≥ 1000 cells/mm3 (1.5 ×109/L)
    2. Platelet count ≥ 100,000 platelet/mm3 (100 ×109/L)
    3. Hemoglobin ≥ 7.5 g/dL.
17. Ability to understand and willingness to sign a written informed consent document.
18. Sexually active participants with female partners of childbearing potential are eligible to participate if they agree to follow 1 of the following methods of contraception consistently, starting from screening, during the study and for at least 3 months after the last dose of ZEN-3694 and/or enzalutamide:

    i. Are abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.

    ii. Are sterilized (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); iii. Agree to use a male condom and have their partner use a contraceptive method with a failure rate of <1% per year as described below when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant, and who agrees to the use of a condom by her partner.

    b. In addition, participants must refrain from donating sperm starting from Screening, during the study and for at least 3 months after the last dose of ZEN-3694 and/or enzalutamide.
19. Sexually active participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse; or use a male condom during each episode of penile penetration during the study
20. Patients with soft-tissue disease amenable to biopsy as determined by Interventional Radiology must agree to serial biopsies as per the study schedule to be eligible.

Exclusion Criteria:

1. Pain due to metastatic prostate cancer requiring treatment intervention with opioid pain medication.
2. ECOG Performance status ≥3
3. Requirement for urinary self-catheterization for voiding due to obstruction secondary to prostatic enlargement well documented to be due to prostate cancer or benign prostatic hyperplasia (BPH). Patients with indwelling Foley or suprapubic catheter for obstructive symptoms are eligible.
4. Active uncontrolled infection. Patients with a history of HIV/AIDS may be eligible if cluster of differentiation 4 (CD4)+ T cell counts are ≥ 350 cell/ul, they have had no opportunistic infection within the past 12 months, they have been on established antiretroviral therapy (ART) for at least four weeks, the HIV viral load is less than 400 copies/ml prior to enrollment, and there is no significant drug-drug interaction with ART and the study drugs. Patients with chronic hepatitis B virus (HBV) infection with active disease who meet criteria for anti HBV therapy are eligible if they are on a suppressive antiviral therapy prior to enrollment and there is no drug-drug interaction with the study drugs. Patients with a history of HCV infection are eligible if they have completed curative antiviral treatment and the hepatitis C virus (HCV) viral load is below the limit of quantification.
5. Any condition or mental impairment that may compromise the ability to give informed consent, patient's safety or compliance with study requirements as determined by the investigator.
6. Patients receiving anticoagulation therapy with warfarin, rivaroxaban, or apixaban are not eligible for study. [Patients on enoxaparin or edoxaban are eligible for study. Patients on warfarin, rivaroxaban, or apixaban, who can be transitioned to one of these alternative agents prior to starting study treatments will be eligible].
7. Patients are excluded with prior history of a thromboembolic event within the last 12 months that are not being treated with systemic anticoagulation.
8. Hematocrit >51%, untreated severe obstructive sleep apnea, uncontrolled or poorly controlled heart failure [per Endocrine Society Clinical Practice Guidelines (34)]
9. Patients allergic to sesame seed oil or cottonseed oil are excluded.
10. Major surgery (i.e. as defined by treating physician) within 3 weeks before screening, or has not fully recovered from prior surgery (i.e., unhealed wound). Note: subjects with planned surgical procedures to be conducted under local anesthesia may participate.

Patients with history of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma, brain arteriovenous malformation).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2031-08-30 (Estimated); Study Completion 2031-08-30 (Estimated)

PRIMARY OUTCOMES:
Clinical/radiographic progression free survival (PFS) with BATZEN | 2 years
  Median time from the first date of BATZEN to the date of first documented radiological progression per RECIST 1.1 for soft tissue or per Prostate Cancer Working Group 3 (PCWG3) for bone lesions, the development of symptoms or complications attributable to cancer progression, or death, whichever occurs first.
Prostate specific antigen (PSA)-Progression free survival (PFS) with ZENZA | 2 years
  PSA-PFS on ZENZA is the median time from start of ZENZA to time of PSA progression according to PCWG3 criteria ,or censored at the last date of PSA assessment for patients without PSA progression.

SECONDARY OUTCOMES:
Number of participants with PSA 50 (≥50% PSA reduction) response to BATZEN | 2 years
  Number of participants with ≥50% PSA reduction from baseline level at screening.
Number of participants with PSA50 response to ZENZA | 2 years
  Number of participants with ≥50% PSA reduction from PSA level at time of progression on BATZEN
Time to PSA progression while on BATZEN | 2 years
  Median time (months) from start of BATZEN to date of PSA progression on ZENZA
Number of participants with Objective response to BATZEN and ZENZA, respectively per RECIST 1.1 criteria | 2 years
  The number of participants with measurable disease who achieve either complete response or partial response to per RECIST 1.1
Progression Free Survival (PFS2) (PSA progression on ZENZA) | 2 years
  Median time from start of BATZEN to date of PSA progression on ZENZA
Overall Survival | 5 years
  Number of months from start of study therapy to death from any cause.
Quality of Life as assessed by the Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Scale | 1 year
  Quality of life over time based on the FACIT-Fatigue. The Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue) is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function. The total score ranges between 0 and 52, with higher scores denoting less fatigue.
Quality of Life as assessed by the Short Form-36 (SF-36) | 1 year
  Quality of life over time based on the SF-36 survey. Short Form 36 (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. Score range 0-100, lower scores represent more physical function disability, while higher scores represent less disability.
Number of participants with treatment-related adverse events | 2 years
  Measured by the number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No